CLINICAL TRIAL: NCT06059430
Title: Cohort Project of Patients With Inflammatory Rheumatism (Rheumatoid Arthritis, Axial and Peripheral Spondyloarthritis Including Psoriatic Arthritis)
Brief Title: Cohort Project of Patients With Inflammatory Rheumatism
Acronym: SMAP
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Rhumato03
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis, Axial; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Axial Spondyloarthritis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — plasma and serum collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient already on treatment: Patients already on biologic or synthetic TRT will be followed for 10 years
  Interventions: Other: no intervention
- Naive patients: Patients who are naive to biological or synthetic treatments
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Chronic inflammatory rheumatism (CIR) is a group of inflammatory diseases that affect the joints and spine and are related to an abnormal immune response. CIR includes many different forms of arthritis that manifest as painful and swollen joints, stiffness, especially in the morning and persisting even after exercise, and limited joint mobility. CIR can also affect bones, cartilage, ligaments, tendons and muscles. Some may affect other organs. These symptoms can lead to a reduced quality of life, limited physical activity and progressive structural and functional deterioration of the joints.

Current treatment for CIR is aimed at reducing inflammation and relieving pain. Anti-inflammatory medications such as corticosteroids and non-steroidal anti-inflammatory drugs can be used to relieve pain and inflammation. Biotherapies can also be used to modify the progression of the disease. On the other hand, regular exercise can help strengthen the muscles that support the affected joints and improve mobility. Physical therapies, such as physical and occupational therapy, can also help improve mobility and relieve pain.

Although there is no definitive cure for CIR early and appropriate treatment can help reduce symptoms and improve quality of life, as well as avoid the risk of developing complications such as lung, cardiovascular, kidney, ophthalmic, liver and other diseases.

It is in this context, in order to better understand CIR to improve the global management of patients, and to analyze the evolution of CIR over time in relation to the different treatments proposed, that the interest in creating a database of patients with CIR arises.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age.
* Patients with rheumatoid arthritis meeting ACR/EULAR criteria or axial and/or peripheral spondyloarthritis meeting ASAS criteria.
* Patients who have failed or are intolerant of DMARDs (methotrexate or arava) for rheumatoid arthritis.
* Patients who have failed treatment with at least two NSAIDs for spondyloarthritis.
* Patients who require biologic/synthetic therapy or patients already receiving biologic or synthetic therapy.

Exclusion Criteria:

- Patient under curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old with rheumatoid arthritis or axial and/or peripheral spondyloarthritis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2043-09-20 (Estimated); Study Completion 2043-12-20 (Estimated)

PRIMARY OUTCOMES:
compare rheumatoid arthritis activity | evrey year during 10 years
  Measurement of disease activity for rheumatoid arthritis using the "Disease Activity Score 28" (DAS28) score ranging from 1 to 6.
compare psoriatic arthritis activity | every year during 10 years
  Measurement of disease activity for psoriatic arthritis using the "Disease Activity Score 44" (DAS44) score ranging from 1 to 6.
compare spondylitis activity | every year during 10 years
  Measurement of disease activity for spondylitis using the "Bath Ankylosing Spondylitis Activity Index" (BASDAI) score ranging from 1 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No